CLINICAL TRIAL: NCT03714971
Title: WhatsApp Embedded in Routine Service Delivery for Smoking Cessation: Effects on Success Rates in a Randomized Controlled Study
Brief Title: WhatsApp Embedded in Routine Service Delivery for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Seyfi Durmaz, PhD MD, research asistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-12.1/11
Record Dates: First submitted 2018-09-04; First posted 2018-10-22 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Smoking Cessation
Keywords: Whatsapp; smoking cessation; cessation service
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: The study was designed as a RCT including two parallel arms: an intervention group receiving messages through WhatsApp Messenger operating on smart phones and a control group not receiving these messages, with an allocation ratio of 1:2. Both groups received the standard outpatient care of the clinic including a 45-60 minutes face-to-face individual counseling at first contact ending with the decision of treatment and quit date, and a support booklet on quitting and subsequent follow-ups by the same clinician at 1st, 2nd, 4th weeks and 3rd month after quit date, either face-to-face at the clinic or by telephone if the patient does not come to the clinic for follow-up. The study was carried out in the smoking cessation clinic of Ege University Medical School's Public Health Department.
Who Masked: Participant, Care Provider
Masking Description: The study was designed as a single-blind study. The physicians (except the first author) were blind to the allocation to intervention or control groups and they conducted their routine smoking cessation counseling work. As long as the patient did not comment on the messages, the physicians were blind throughout the follow ups as well. After the first routine counseling, participants were informed by the first author about the study, thus they were not blind to the intervention. The analysis of the study was conducted by the first author who was not blind to the intervention/ control status of the participants. The first author could not be blind as he was to send out the WhatssApp messages. However, contact numbers of the participants were labeled with numbers (I-01 to I-44) to secure anonymity and to prevent any bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving WhatsApp messages (Experimental): Among patients applying to the smoking cessation outpatient clinic between March and October 2017, >18-year old volunteers who smoked at least one cigarette/day, using WhatsApp at least on four days of the week, accepting the 3-month follow-up were included In receiving WhatsApp messages group.
  Interventions: Behavioral: WhatsApp embedded in smoking cessation service
- Not receiving WhatsApp messages (No Intervention): In "not receiving WhatsApp messages" group; Stratification and randomization were both used to randomly allocate participants to both arms of the study. The intervention and control groups were first stratified according to physician and then gender, and later allocated in a simple random manner. Randomization was conducted using a computer spreadsheet. Allocation according to gender was conducted regarding the 2:3 female to male ratio in the routine cessation services and stratification according to physician aimed to have a balanced distribution among the different physicians working in the same cessation unit. As the target number of participants was small, further stratification was not applied. Simple random sampling was then used to allocate participants to each group.

INTERVENTIONS:
Behavioral: WhatsApp embedded in smoking cessation service — The routine service delivery was ongoing as the intervention was conducted. In addition to the routine procedures in service delivery described above, WhatsApp messages were sent according to the plan.
  Arms: Receiving WhatsApp messages

SUMMARY:
Background: Recently, the use of communication technologies and social media applications has become increasingly widespread to strengthen efforts for smoking cessation. The purpose of this study is; to assess the effect on success rate of the WhatsApp application which is embedded in the smoking cessation policlinic service delivery.

Materials and Methods: A randomized controlled intervention study was conducted with 132 volunteers who were followed up at the EUTF Smoking Cessation Policlinic between March-July 2017. The intervention content based on transtheoretic model was prepared and 60 WhatsApp messages were delivered to participants for 3 months of follow up. For data collection, initial interview form and follow up form consisting sociodemographic characteristics, smoking status, medical condition and treatment, were used. The success rate at first and third months were assessed by the point-prevalence regarding the previous week. Intention-to-treat analysis was used. For secondary outcomes; number of follow-ups, change in weight and continuity of medication were evaluated.

Findings: Success rate in the first month was 65.9% for intervention group and 40.9% in the control group; for the third month it was 50.0% in the intervention group and 30.7% in the control group. Being in the intervention group increased the success rate by 3,50 (1,30-9,44) times in the first month and 2,50 (1,08-6,40) times in the third month. The intervention was the only parameter effective in the two follow-up periods; the difference in success rate caused by gender, marital status and work-related social class has been eliminated after adjustment for the intervention.

DETAILED DESCRIPTION:
Trial design

The study was designed as a RCT including two parallel arms: an intervention group receiving messages through WhatsApp Messenger operating on smart phones and a control group not receiving these messages. Both groups received the standard outpatient care of the clinic including aproximately 45 minutes face-to-face individual counseling at first contact ending with the decision of treatment and quit date, and a support booklet on quitting and subsequent follow-ups by the same clinician at 1st, 2nd, 4th weeks and 3rd month after quit date, either face-to-face at the clinic or by telephone if the patient does not come to the clinic for follow-up. The study was carried out in the smoking cessation clinic of Ege University Medical School's Public Health Department.

Sample size

An a priori power analysis was conducted with OpenEpi, Version 3 by selecting a two-sided test to compare 30% success in the control group at 1st month versus 60% success rate in the intervention group with an error margin of 5%, a power of 80% and an allocation ratio of 1:2 which yielded a minimum sample size of 36 in the intervention and 72 in the control groups. For possible loss to follow-up, the sample sizes were increased by 20% to 43 and 86, respectively.

Randomization

Among the 132 participants included in the study, 44 were randomly allocated to the intervention arm and 88 were randomly allocated to the control group. Among the intervention group , there were no losses to follow-up at 1st and 3rd months, but two participants have requested the cessation of the intervention after their 1st month follow-up.

Blinding

The study was single-blind as blinding of the helthcare providers to intervention assignment was achieved and the physicians conducted usual care for smoking cessation counseling.The physicians were blind throughout the follow ups as well. However, participants and the researcher who sent the messages were not blind.

Variables

Primary outcome variables: Quitting success rates at the end of the 1st, 3rd and 6th month of follow-up in the intervention and control groups. Quitting success rate at 1st month was calculated with point prevalence. History of cessation was based on self report and those who declared not smoked even a single puff on a cigarette at all in the past two weeks were considered as "successful" in the quitting attempt. The success rate at 3rd month was calculated with point prevalence. In this point, not smoking at all in total in the past ten weeks was considered "successful" in the quitting attempt. The success rate at 6th month was calculated with point prevalence. In this point, not smoking at all in total in the past 24 weeks was considered "successful" in the quitting attempt.

Secondary outcome variables: The total number of follow-ups in the 1st, 3rd and 6th month. Contacts were divided into two categories: face-to face contacts and telephone calls. The total number of routine follow-ups was classified as adequate when 3 or more in the 1st month and a total of 4 follow-ups was considered as adequate at 3rd month. At 1st month, at least one of these follow-ups was required to be face-to-face for adequacy. The continuity to drug/NRT therapy was categorized as <1 month or ≥1 month. Any change in weight was categorized as; has weight gain, no weight gain

Data collection Data collection was conducted at the Smoking Cessation Clinic of the Public Health Department at Ege University Medical School Hospital between March 2017-March 2018. The intended number of participants was achieved in 4.5 months and with the completion of the last follow-up, the study was finalized.

Analysis

The analyses were conducted according to the Intention-To-Treat (ITT) principle. The participants lost to follow-up were considered unsuccessful in quitting, as non-response could be expected in relapsing individuals, thus Last Observation Carried Forward (LOCF) was not used.

Smoking cessation successes in the groups were compared with the incidences and relative efficacy of the intervention. Chi-square test, Student's t test in independent groups, single and multivariate logistic regression (enter method) were used for analyses. The multivariate analysis of factors associated with smoking cessation success was performed by using logistic regression analysis with two models. In the first model the investigators controlled for age and gender, in the second model controlling was for age, gender and all the other associated variables in univariate analyses. Analyses were made separately for the 1st, 3rd and 6th month. Statistical significance was set at p<0.05.

Ethical issues

The study was approved by Ege University Medical School's institutional review board (decision no.16-12.1/11 on January 6, 2017). Written informed consent of every participant to enroll and receive WhatsApp messages were also obtained with confidentiality for name and address. With the blinding procedures described above, the delivery of routine service for all participants regardless of the allocation to intervention or control group was ensured.

ELIGIBILITY:
Inclusion Criteria:

* Among patients applying to the smoking cessation outpatient clinic between March and October 2017,
* >18-year old volunteers who smoked at least one cigarette/day,
* using WhatsApp at least on four days of the week,
* accepting the 3-month follow-up were included in the study.

Exclusion Criteria:

* Besides people who did not meet the inclusion criteria, other patients applying to the clinic but who were referred to another centre without receiving any treatment,
* people who were not 'ready to quit' according to the TTM stages of change evaluation
* who had already quit before applying to the clinic were excluded.
* If two or more patients were living in the same house or had applied to the clinic together, only the first of these was included and the rest were excluded from the study, as they could show the arriving messages to their friend/ partner/ relative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Quitting success rates at the end of the 1st, 3rd and 6th month | 6 months
  Quitting success rates at the end of the 1st, 3rd and 6th month of follow-up in the intervention and control groups. Quitting success rate at 1st month was calculated with point prevalence. History of cessation was based on self report and those who declared not smoked even a single puff on a cigarette at all in the past two weeks were considered as "successful" in the quitting attempt (19). The success rate at 3rd month was calculated with point prevalence. In this point, not smoking at all in total in the past ten weeks was considered "successful" in the quitting attempt. The success rate at 6th month was calculated with point prevalence. In this point, not smoking at all in total in the past 24 weeks was considered "successful" in the quitting attempt.
  A decrease in success rates at six months is expected in comparison with 3 months as the intervention lasts for 3 months.

SECONDARY OUTCOMES:
The total number of follow-ups | 3 months
  The total number of follow-ups in the 1st, 3rd month. Contacts were divided into two categories: face-to face contacts and telephone calls. The total number of routine follow-ups was classified as adequate when 3 or more in the 1st month and a total of 4 follow-ups was considered as adequate at 3rd month. At 1st month, at least one of these follow-ups was required to be face-to-face for adequacy.
The continuity to drug, | 3 months
  The continuity to drug/NRT therapy was categorized as using the prescribed drug for <1 month or ≥1 month.
Self reported difference in weight in kilograms since the first contact | 3 months
  Any increase in weight (kg) was categorized as; has weight gain, no weight gain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Nedicine Public Health Departmant, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filozof C, Fernandez Pinilla MC, Fernandez-Cruz A. Smoking cessation and weight gain. Obes Rev. 2004 May;5(2):95-103. doi: 10.1111/j.1467-789X.2004.00131.x. PMID 15086863
- [Background] Munoz RF, Chen K, Bunge EL, Bravin JI, Shaughnessy EA, Perez-Stable EJ. Reaching Spanish-speaking smokers online: a 10-year worldwide research program. Rev Panam Salud Publica. 2014 May-Jun;35(5-6):407-14. PMID 25211569
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Cheung YT, Chan CH, Lai CK, Chan WF, Wang MP, Li HC, Chan SS, Lam TH. Using WhatsApp and Facebook Online Social Groups for Smoking Relapse Prevention for Recent Quitters: A Pilot Pragmatic Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Oct 22;17(10):e238. doi: 10.2196/jmir.4829. PMID 26494159
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Apr 10;4(4):CD006611. doi: 10.1002/14651858.CD006611.pub4. PMID 27060875
- [Background] Carlson LE, Goodey E, Bennett MH, Taenzer P, Koopmans J. The addition of social support to a community-based large-group behavioral smoking cessation intervention: improved cessation rates and gender differences. Addict Behav. 2002 Jul-Aug;27(4):547-59. doi: 10.1016/s0306-4603(01)00192-7. PMID 12188591
- [Background] Turner J, McNeill A, Coleman T, Bee JL, Agboola S. Feasibility of offering nicotine replacement therapy as a relapse prevention treatment in routine smoking cessation services. BMC Health Serv Res. 2013 Feb 1;13:38. doi: 10.1186/1472-6963-13-38. PMID 23375024
- [Derived] Durmaz S, Ergin I, Durusoy R, Hassoy H, Caliskan A, Okyay P. WhatsApp embedded in routine service delivery for smoking cessation: effects on abstinence rates in a randomized controlled study. BMC Public Health. 2019 Apr 8;19(1):387. doi: 10.1186/s12889-019-6727-z. PMID 30961557
- See also: WHO report on the global tobacco epidemic, 2017: monitoring tobacco use and prevention policies — http://apps.who.int/iris/handle/10665/255874
- See also: WhatsApp: number of users 2013-2017 — https://www.statista.com/statistics/260819/number-of-monthly-active-whatsapp-users/